CLINICAL TRIAL: NCT03214302
Title: The Incidence of Postpartum Hepatitis in Pregnant Women With High HBVDNA Loads
Brief Title: The Incidence of Postpartum Hepatitis in Pregnant Women With Chronic Hepatitis B Virus Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XMLX201706-2
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis B
Keywords: antiviral treatment; hepatitis B virus; pregnant woman; Postpartum hepatitis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- control group (No Intervention): In this group, pregnant women with HBsAg/HBeAg positive and HBV DNA > 106 copies/ml don not use any antiviral drugs during pregnancy.healthy Pregnant women with HBsAg(-), HBeAg(-)
- experimental group (Experimental): pregnant women with HBsAg/HBeAg positive and HBV DNA > 106 copies/ml start to use Tenofovir Disoproxil Fumarate(TDF) antiviral treatment from the 32 weeks of gestation and drug withdrawal after delivery immediately, and drug withdrawal in the 6 weeks after delivery.
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Tenofovir Disoproxil Fumarate was used for the experimental group of pregnancy women in the 32 weeks during pregnancy
  Other Names: TDF
  Arms: experimental group

SUMMARY:
The majority of childbearing age women with hepatitis B virus infection were still in the immune tolerance period. Our recent research had shown that most puerperae after delivery had elevated ALT level. However, there is no withdrawal time recommendations after childbirth at present.Through the study of hepatitis occurrence after delivery and drug withdrawal, the investigators explore the withdrawal time of antiviral treatment during pregnancy.

DETAILED DESCRIPTION:
Most of childbearing age women with hepatitis B virus infection were still in the immune tolerance period. Our recent research had shown that most puerperae after delivery had elevated ALT level, and 11.5% of patients with HBV DNA positive would lead to deterioration of liver function. Meanwhile, the highest peak of ALT level could occur in 2 weeks after delivery, then it would dropped to a low point in 4-5 weeks. However, there is no withdrawal time recommendations after childbirth at present.The aim of our study is to investigate the changes of serological indexes, the changing rule of the liver function, hepatitis status, and its correlation with antiviral therapy in pregnant women with HBV infection after delivery, and then explore the withdrawal time of antiviral treatment during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were chronic hepatitis B and had achieved HBeAg positive and HBV DNA > 106 copies/ml
* healthy Pregnant women with HBsAg(-), HBeAg(-)

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus, HIV, etc.
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver
* without gestational hypertension, premature rupture of membranes, antepartum haemorrhage diseases or amniotic fluid piercing history during pregnancy.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 560 (Estimated)
Dates: Start 2017-01-01; Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of hepatitis flare after drug withdrawal in maternal postpartum | after delivery 24weeks
  ALT > 3 times the upper limit of normal

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li M, Sun F, Bi X, Lin Y, Yang L, Jiang T, Deng W, Lu Y, Zhang L, Yi W, Xie Y. Effects of antiviral therapy and drug withdrawal on postpartum hepatitis in pregnant women with chronic HBV infection. Hepatol Int. 2023 Feb;17(1):42-51. doi: 10.1007/s12072-022-10412-w. Epub 2022 Sep 15. PMID 36109430
- [Derived] Wang F, Xie S, Ran C, Hao H, Jiang T, Deng W, Bi X, Lin Y, Yang L, Sun F, Zeng Z, Xie Y, Li M, Yi W. Effect of Antiviral Therapy During Pregnancy on Natural Killer Cells in Pregnant Women With Chronic HBV Infection. Front Immunol. 2022 May 23;13:893628. doi: 10.3389/fimmu.2022.893628. eCollection 2022. PMID 35677040